CLINICAL TRIAL: NCT02368080
Title: Multiple Breath Nitrogen Washout in Healthy and Cystic Fibrosis Adults: a Comparison of Two Commercially Available Devices
Brief Title: Multiple Breath Nitrogen Washout in Healthy and Cystic Fibrosis Adults
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Poncin, Physiotherapist, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: StLuc MBWN2 01
Record Dates: First submitted 2015-01-14; First posted 2015-02-20 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Cystic Fibrosis; Healthy
Keywords: Lung Clearance Index; Cystic Fibrosis; Multiple Breath Nitrogen Washout
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cystic fibrosis adults (CF): No treatment, comparison of LCI values obtained with two devices
  Interventions: Device: Comparison of two MBWN2 devices : "EasyOne Pro Lab" versus "Exhalyzer D"
- Healthy adults (HC): No treatment, comparison of LCI values obtained with two devices Free of respiratory disease or others diseases likely to disturb respiratory system.
  Interventions: Device: Comparison of two MBWN2 devices : "EasyOne Pro Lab" versus "Exhalyzer D"

INTERVENTIONS:
Device: Comparison of two MBWN2 devices : "EasyOne Pro Lab" versus "Exhalyzer D" — Healthy and Cystic Fibrosis participants will perform the same day MBWN2 tests in duplicate with each device.

SUMMARY:
This study compares the lung clearance index (LCI) in cystic fibrosis and healthy adults obtained with two different multiple breath nitrogen washout (MBWN2) devices. Each participants will perform the test (LCI) in duplicate on each device.

DETAILED DESCRIPTION:
Using nitrogen as the inert gas, there are currently two commercially available devices that offer the possibility to measure the LCI. However, comparison between them are lacking. The 2 MBWN2 devices are the "EasyOne Pro Lab" (ndd Medical Technologies, Zürich, Switzerland) and the "Exhalyzer D" (Eco Medics AG, Duernten, Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis diagnosis

Exclusion Criteria:

* Respiratory infection within 3 weeks
* Chronically infected with methicillin-resistant Staphylococcus aureus or Burkholderia Cepacia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CF : primary care clinic HC : community sample
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Lung Clearance Index (LCI) | 1 hour

SECONDARY OUTCOMES:
Discriminative ability of LCI of each device (assessed by evaluating the proportion of patients with normal spirometry but high LCI with each device) | 1 hour
  Difference in discriminative ability between devices will be assessed by evaluating the proportion of patients with normal spirometry but high LCI with each device
Functional residual capacity (FRC) ( the helium rebreathing technique (FRC He) with a "Jaeger Masterscreen" (Würzburg, Germany) | 1 hour
  FRC will be compared with a third device in a subset of 11 healthy adults : the helium rebreathing technique (FRC He) with a "Jaeger Masterscreen" (Würzburg, Germany)

OTHER OUTCOMES:
Subject's preference | 1 hour
  Just after the completion of the tests, subjects will be asked to answer which one of the device they most preferred (i.e.: device A or device B or no preference).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Lebecque, MD, PhD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; William Poncin, PhD student, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Anne-Sophie Aubriot, PhD student, Study Chair — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium